CLINICAL TRIAL: NCT03335982
Title: Feasibility and Safety of Ttransendoscopic Enteral Tubing in Mid-gut
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Second Hospital of Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Faming Zhang, Associate professor, Gastroenterology, The Second Hospital of Nanjing Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: TET-CN-151001
Record Dates: First submitted 2017-10-27; First posted 2017-11-08 (Actual); Last update posted 2017-12-02 (Actual); Status verified 2017-09

CONDITIONS: Transendoscopic Enteral Tubing
Keywords: transendoscopic enteral tubing; mid-gut; endoscopy; nasal-jejunal tube; fecal microbiota transplantation; enteral nutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- transendoscopic enteral tubing in mid-gut (Other): A TET tube was inserted into mid-gut through the nasal orifice and fixed on the pylorus wall by one tiny titanium endoscopic clip under anesthesia. The feasibility, safety, success rate, and satisfaction with TET placement were evaluated for enteral nutrition or fecal microbiota transplantation.
  Interventions: Procedure: transendoscopic enteral tubing in mid-gut

INTERVENTIONS:
Procedure: transendoscopic enteral tubing in mid-gut — A TET tube was inserted into mid-gut through the nasal orifice and fixed on the pylorus wall by one tiny titanium endoscopic clip under anesthesia.

SUMMARY:
A transendoscopic enteral tubing (TET ) tube was inserted into mid-gut through the nasal orifice and fixed on the pylorus wall by one tiny titanium endoscopic clip under anesthesia. This study aimed to evaluate the feasibility and safety of TET in mid-gut .

DETAILED DESCRIPTION:
In recent years, fecal microbiota transplantation (FMT) has gained appeal as a therapeutic option worldwide. Traditionally, microbiota can be administered through the upper-gut, the mid-gut, and the lower-gut pathways. FMT via colonoscopy is a classic approach, but in our previous study on ulcerative colitis, those patients have difficulty to maintain the infused microbiota suspension for enough time through this way. Thus, the investigators designed the colonic transendoscopic enteral tubing (TET) technology, which made whole-colon administration of treatment and repeat FMTs possible. However, some patients are resistant to undergo bowel preparation for colonoscopy or some are not suitable for colonic delivering way. Therefore, mid-gut delivering way is an important option for those patients. In previous researches on FMT for Crohn's disease, patients and physician faced the similar problem that some patients need repeat FMT during hospitalization, and some may need enteral nutrition at the same time. In order to have a quicker and more convenient placement of mid-gut/nasal-jejunal TET tube than traditional methods, the investigators designed a novel mid-gut TET technique without further confirmation for the location of tube in gut by X-ray or other medical devices after the endoscopic procedure. This study aimed to evaluate the feasibility, safety, and value of the mid-gut TET technique.

ELIGIBILITY:
Inclusion Criteria:

Mild to moderate inflammatory bowel disease (Montreal classification) or suitability for endoscopy, and consented to undergo TET placement for their diseases and conditions

Exclusion Criteria:

No history of using Biologic, immunomodulatory therapy or corticosteroid therapy.

With contraindication of endoscopy. Pregnant or lactating female

Ages: 5 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-08-01 (Actual); Primary Completion 2017-12-01 (Estimated); Study Completion 2017-12-01 (Estimated)

PRIMARY OUTCOMES:
success rate | All patients were followed up from date of intubation to one mouth after discharge
  the success rate of of the TET procedure
adverse events rate | All patients were followed up from date of intubation to one mouth after discharge
  Procedure-related and tube-related adverse events after procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Medical Center for Digestive Diseases, The Second Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Cui B, Feng Q, Wang H, Wang M, Peng Z, Li P, Huang G, Liu Z, Wu P, Fan Z, Ji G, Wang X, Wu K, Fan D, Zhang F. Fecal microbiota transplantation through mid-gut for refractory Crohn's disease: safety, feasibility, and efficacy trial results. J Gastroenterol Hepatol. 2015 Jan;30(1):51-8. doi: 10.1111/jgh.12727. PMID 25168749
- [Background] Cui B, Li P, Xu L, Zhao Y, Wang H, Peng Z, Xu H, Xiang J, He Z, Zhang T, Nie Y, Wu K, Fan D, Ji G, Zhang F. Step-up fecal microbiota transplantation strategy: a pilot study for steroid-dependent ulcerative colitis. J Transl Med. 2015 Sep 12;13:298. doi: 10.1186/s12967-015-0646-2. PMID 26363929
- [Background] Peng Z, Xiang J, He Z, Zhang T, Xu L, Cui B, Li P, Huang G, Ji G, Nie Y, Wu K, Fan D, Zhang F. Colonic transendoscopic enteral tubing: A novel way of transplanting fecal microbiota. Endosc Int Open. 2016 Jun;4(6):E610-3. doi: 10.1055/s-0042-105205. Epub 2016 Apr 28. PMID 27556065